CLINICAL TRIAL: NCT02192099
Title: Phase 2, Open Label Extension for Subjects With Inadequate/Partial Response to Antidepressants During the Current Episode of Major Depressive Disorder Previously Treated With GLYX-13 (Extension of GLYX13-C-202, NCT01684163)
Brief Title: Open Label Extension for GLYX13-C-202, NCT01684163
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Patients from this study were rolled into RAP-MD-99.
Sponsor: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLYX13-C-203
Record Dates: First submitted 2014-07-08; First posted 2014-07-16 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — GLYX-13 peptide; Organization and Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rapastinel (225 mg/450 mg IV administration) prefilled syringe (Experimental): Investigators began treatment in RAP-MD-05 based on the dose level to which the patient was assigned during participation in GLYX13-C-202; patients originally assigned to rapastinel 5 mg/kg received rapastinel 225 mg, and patients originally assigned to rapastinel 10 mg/kg received rapastinel 450 mg. Investigators had the option to decrease the dose level from 450 to 225 mg if a patient experienced an adverse event(s) that the investigator believed may be associated with rapastinel
  Interventions: Drug: Rapastinel (225 mg/450 mg IV administration)

INTERVENTIONS:
Drug: Rapastinel (225 mg/450 mg IV administration) — Investigators began treatment in RAP-MD-05 based on the dose level to which the patient was assigned during participation in GLYX13-C-202; patients originally assigned to rapastinel 5 mg/kg received rapastinel 225 mg, and patients originally assigned to rapastinel 10 mg/kg received rapastinel 450 mg. Investigators had the option to decrease the dose level from 450 to 225 mg if a patient experienced an adverse event(s) that the investigator believed may be associated with rapastinel
  Other Names: GLYX-13 IV Dose

SUMMARY:
Examine the safety of long term repeat exposure to GLYX-13 in subjects who participated in GLYX13-C-202.

DETAILED DESCRIPTION:
Examine the safety of long term repeat exposure to GLYX-13 in subjects who participated in GLYX13-C-202 in an open label extension trial.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have completed 8 weeks of treatment in the preceding study (GLYX13-C-202, NCT01684163.
2. Participants who wish to continue treatment with GLYX-13 after the preceding study.
3. Meets Diagnostic and Statistical Manual, Fourth Edition, Text Revision (DSM-IV-TR) criteria for major depressive disorder (MDD).
4. Female subjects of childbearing potential with a negative serum pregnancy test prior to entry into the study and who are practicing an adequate method of birth control (eg oral or parenteral contraceptives, intrauterine device, barrier, abstinence) and who do not plan to become pregnant during the course of the study. Female subjects may be included without a negative serum pregnancy test if they are surgically sterile or at least 2 years post-menopausal.
5. Clinical laboratory values <2 times the upper limit of normal (ULN) or deemed not clinically significant per the investigator and Naurex medical monitor.
6. Ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments.
7. Based on the investigator and Naurex medical monitor's clinical judgment, subjects with eating disorders, obsessive compulsive disorder (OCD), panic disorder, post-traumatic stress disorder (PTSD), and generalized anxiety disorders secondary to major depressive episodes (MDEs) are permitted.

Exclusion Criteria:

1. Axis I diagnosis of delirium, dementia, dysthymia, amnestic or other cognitive disorder, schizophrenia or other psychotic disorder, bipolar I or II disorder, eating disorder (anorexia or bulimia nervosa), obsessive-compulsive disorder, panic disorder, acute stress disorder, agoraphobia, social phobia, attention-deficit hyperactivity disorder (ADHD), or PTSD.
2. A clinically significant current Axis II diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal, or histrionic personality disorder
3. Experiencing hallucinations, delusions, or any psychotic symptomatology in the current episode; lifetime history of psychosis.
4. Huntington's, Parkinson's, Alzheimer's, Multiple Sclerosis, or a history of seizures or strokes.
5. Currently hospitalized or residing in an in-patient facility during study participation.
6. Substance abuse since the end of participation in GLYX13-C-202, including greater than or equal to 5 units of alcohol per day where 1 unit = ½ pint of beer, 1 glass of wine 4 oz, or 1 oz. of spirits consumed most weeks or in the opinion of the investigator
7. Women who are planning to become pregnant during the course of the study.
8. Allergy or intolerance to current antidepressant or other current medications.
9. Participation in any clinical trial of an investigational product or device within 30 days of enrollment in this trial with the exception of GLYX13-C-202.
10. Positive screen for drugs of abuse: cocaine, marijuana, PCP, ketamine, opioid or other agent that in the opinion of the investigator is being abused
11. Pose current (past 6 months) suicide risk based on administration of the C SSRS and the investigator's clinical judgment.
12. Human immunodeficiency virus (HIV) infection (based on the based on the HIV-1 & HIV-2 antibody screen) or other ongoing infectious disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-09-08 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Hoogerheyde, Study Director — Allergan
Locations (10):
- United States (10):
  - Office of Psychiatric Research, Birmingham, Alabama
  - Artemis Institute for Clinical Research, San Diego, California
  - Chicago Research Center, Chicago, Illinois
  - University of Kansas School of Medicine Clinical Trial Unit, Wichita, Kansas
  - PharmaSite Research, Inc., Baltimore, Maryland
  - Boston Clinical Trials Inc., Roslindale, Massachusetts
  - Woodlands Professional Princeton Medical Institute Building, Princeton, New Jersey
  - Finger Lake Clinical Research, Rochester, New York
  - Lindner Center of HOPE, Mason, Ohio
  - PRA Health Sciences Phase 2/3 Outpatient & CNS Clinic, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Outpatients who have completed 8 or more weeks of treatment in the preceding study (GLYX13-C-202) and were willing to continue treatment with rapastinel (GLYX-13). Patients originally assigned to rapastinel 5 mg/kg received rapastinel 225 mg, and patients originally assigned to rapastinel 10 mg/kg received rapastinel 450 mg.
Groups:
- Rapastinel (GLYX-13) 225mg or 450 mg IV Administration: Rapastinel (225 mg/450 mg intravenous [IV] administration), prefilled syringe.
Period: Overall Study
Arm/Group | Rapastinel (GLYX-13) 225mg or 450 mg IV Administration
Started | 61
Completed | 0
Not Completed | 61
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 1
Not completed — Pregnancy | 1
Not completed — Protocol Violation | 8
Not completed — Study Terminated by Sponsor | 32
Not completed — Withdrawal by Subject | 11
Not completed — Miscellaneous Reasons | 5

BASELINE CHARACTERISTICS:
Population: The Safety Population will consist of all subjects who received any injection of study drug.
Arm/Group | Rapastinel (GLYX-13) 225mg or 450 mg IV Administration
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.4 (10.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 57
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 48
  Black or African American | 13

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Experience an Adverse Event Over the Course of the Study.
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. A TEAE was an AE that occurred after receiving the first dose of investigational product or an AE present prior to first dose but increased in severity during the Treatment Period.
Time Frame: 48 Months
Population: The Safety Population will consist of all subjects who received any injection of study drug.
Measure: Number; unit: Participants
Arm/Group | Rapastinel (GLYX-13) 225mg or 450 mg IV Administration
Number analyzed (Participants) | 61
Participants | 60

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for up to 48 months.
Description: The Safety Population will consist of all subjects who received any injection of study drug.
Arm/Group | Rapastinel (GLYX-13) 225mg or 450 mg IV Administration
All-Cause Mortality (participants affected / at risk) | 0/61
Serious Adverse Events (participants affected / at risk) | 14/61
Other Adverse Events (participants affected / at risk) | 60/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rapastinel (GLYX-13) 225mg or 450 mg IV Administration (N=61)
Drug use disorder (Psychiatric disorders) | 2
Seizure (Nervous system disorders) | 2
Appendicitis (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Colitis (Gastrointestinal disorders) | 1
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1
Depression (Psychiatric disorders) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hemiparesis (Nervous system disorders) | 1
Lacunar stroke (Nervous system disorders) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Ureteric injury (Injury, poisoning and procedural complications) | 1
Volvulus of small bowel (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Rapastinel (GLYX-13) 225mg or 450 mg IV Administration (N=61)
Upper respiratory tract infection (Infections and infestations) | 33
Headache (Nervous system disorders) | 31
Diarrhoea (Gastrointestinal disorders) | 28
Nausea (Gastrointestinal disorders) | 24
Back pain (Musculoskeletal and connective tissue disorders) | 16
Viral upper respiratory tract infection (Infections and infestations) | 16
Insomnia (Psychiatric disorders) | 14
Vomiting (Gastrointestinal disorders) | 13
Anxiety (Psychiatric disorders) | 12
Constipation (Gastrointestinal disorders) | 12
Abdominal pain (Gastrointestinal disorders) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Sinusitis (Infections and infestations) | 11
Gastroenteritis (Infections and infestations) | 10
Influenza (Infections and infestations) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10
Fatigue (General disorders) | 9
Abdominal pain upper (Gastrointestinal disorders) | 8
Depression (Psychiatric disorders) | 8
Dry mouth (Gastrointestinal disorders) | 8
Dizziness (Nervous system disorders) | 7
Electrocardiogram QT prolonged (Investigations) | 6
Ligament sprain (Injury, poisoning and procedural complications) | 7
Migraine (Nervous system disorders) | 7
Hypoaesthesia (Nervous system disorders) | 6
Irritability (Psychiatric disorders) | 6
Muscle strain (Injury, poisoning and procedural complications) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Pharyngitis (Infections and infestations) | 6
Weight increased (Investigations) | 6
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 5
Blood pressure increased (Investigations) | 5
Bronchitis (Infections and infestations) | 5
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Pollakiuria (Renal and urinary disorders) | 5
Procedural pain (Injury, poisoning and procedural complications) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Toothache (Gastrointestinal disorders) | 5
Urinary tract infection (Infections and infestations) | 5
Vertigo (Ear and labyrinth disorders) | 5
Arthropod bite (Injury, poisoning and procedural complications) | 4
Decreased appetite (Metabolism and nutrition disorders) | 4
Ear infection (Infections and infestations) | 4
Eye irritation (Eye disorders) | 4
Fall (Injury, poisoning and procedural complications) | 4
Hypertension (Vascular disorders) | 4
Increased appetite (Metabolism and nutrition disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Oedema peripheral (General disorders) | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 4
Seasonal allergy (Immune system disorders) | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4
Skin abrasion (Injury, poisoning and procedural complications) | 4
Weight decreased (Investigations) | 4
Vulvovaginal mycotic infection (Infections and infestations) | 3/46
Erectile dysfunction (Reproductive system and breast disorders) | 1/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-11-23): https://cdn.clinicaltrials.gov/large-docs/99/NCT02192099/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT02192099/SAP_001.pdf